CLINICAL TRIAL: NCT02999386
Title: Role Of Stress Induced Hyperglycemia On The Outcome Of Trauma Patients
Brief Title: Stress Induced Hyperglycemia In Trauma
Acronym: SIHG
Status: Completed | Type: Observational
Sponsor: Hamad Medical Corporation (Industry)
Responsible Party: Principal Investigator, Dr. Ayman El-Menyar, Associate Professor, Hamad Medical Corporation
Other Study IDs: 14471/14
Record Dates: First submitted 2016-12-15; First posted 2016-12-21 (Estimated); Last update posted 2020-07-23 (Actual); Status verified 2020-07

CONDITIONS: Trauma; Stress Induced Hyperglycemia; Diabetes Mellitus
Keywords: stress, hyperglycemia, inflammatory markers, trauma, HbA1c; interleukin-6
MeSH Terms: conditions — Wounds and Injuries; Diabetes Mellitus; Hyperglycemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The clinical relevance of the observed stress induced hyperglycemia in trauma patients remains unclear. The earlier studies suggested the implications of cytokines in stress induced hyperglycemia and the outcomes after trauma. To date, there is little information available regarding the effect of diabetic hyperglycemia (occult or known) on outcomes after trauma and whether these patients represent a distinct group with differential outcomes when compared to those with stress-induced hyperglycemia. Herein, the purpose of this study is to identify the incidence of stress induced hyperglycemia as well as diabetic hyperglycemia in trauma patients and to investigate the association between proinflammatory cytokine levels and hyperglycemia in our trauma population.

DETAILED DESCRIPTION:
Intensive glucose control is vital for prognosis and preservation of normal physiologic status in trauma patients. The acute effects of severe trauma, infection, and surgery result in remarkable metabolic stress on the human body. Hyperglycemia is a normal metabolic response to stress and injury [1]. Irrespective of the involved injury mechanism, post-traumatic metabolic changes occur due to stress in terms of an increased glucose production, decreased insulin production, and insulin resistance in the peripheral tissues and eventually lead to a state of hyperglycemia. Traumatic injury also induces changes in endogenous hormone production and enhanced utilization of metabolites that usually lead to stress related hyperglycemia. Measurement of HbA1c levels can be used as a screening tool to discriminate unknown diabetes mellitus from stress-induced hyperglycemia (SIH). Published studies that have evaluated the association between presenting hyperglycemia and worse outcomes in trauma patients have all consistently showed higher mortality and infection rates in patients presented with elevated serum glucose levels of 200 mg/dL or more [2-5]. A recent study evaluated the differential effect of SIH in comparison to diabetic hyperglycemia (DH) on outcomes in trauma victims. The authors observed that as opposed to DH, SIH is associated with a higher mortality rate after injury [4]. A prospective study of patients with severe traumatic brain injury demonstrated that admission glucose levels >11.1 mmol/L were associated with increased mortality and poor neurologic outcomes [6]. Stress associated with critical illness is characterized by the activation of inflammatory cellular mediators [7]. During acute illness there is an increase in the systemic inflammatory response that is characterized by increased production of pro-inflammatory cytokines. Importantly, there is relationship between abnormal cytokine production and hyperglycemia in severe sepsis patients which aggravates the immune response leading to poor clinical outcomes. Recent studies suggested that interleukin-6 (IL-6) is involved in glucose metabolism and insulin action. The proinflammatory IL-6 is normally released upon infection; however, it induces insulin resistance during conditions of hyperglycemia [8]. Moreover, IL-18 levels are significantly elevated in diabetic patients with microalbuminuria as compared with patients with normoalbuminuria [9]. This might indicate that certain interleukins (IL) are involved in the pathogenesis of SIH. Though, the clinical relevance of the observed SIH in trauma patients remains unclear. The earlier studies suggested the implications of cytokines in SIH and outcomes after trauma. To date, there is little information regarding the effect of diabetic hyperglycemia (occult or known) on the clinical outcomes after trauma and whether these patients represent a distinct group with differential outcomes when compared to those with SIH. The purpose of this study is to identify the incidence of SIH as well as diabetic hyperglycemia in trauma patients and to investigate the association between the proinflammatory cytokine levels and hyperglycemia in trauma population.

Primary objective:

- To evaluate the outcomes of stress induced hyperglycemia in patients presented with traumatic injury.

Secondary objectives:

* To investigate the association between pro-inflammatory cytokine levels and SIH in trauma patients.
* To identify the incidence of SIH and occult diabetes mellitus in trauma population.

It is a prospective study which will include all adult trauma patients who require hospital admission and have been investigated for random plasma glucose level and HbA1C measured within 5 hours of admission. All trauma patients will undergo thorough clinical assessment and resuscitation according to the Advanced Trauma Life Support (ATLS) guidelines. The present study will screen all traumatic injury patients presented to the trauma room and those who are willing to participate and provide written informed consent or consented by the relatives or used emergency consent (Exception from Informed Consent Requirements for Emergency Research" Policy # 11026) to draw blood for the investigations will be included in the study. All the study subjects will be managed according to the standard care of the hospital. The investigators will directly access all adult traumatic injury patients that will be presented to the trauma room and review the medical file and/or electronic medical record (EMR) to confirm the eligibility. Usually trauma patients are unconscious, under shock and are physically and mentally unfit to communicate or sign consent. The trauma surgeon will explain the consent form to the legal representatives of the subjects in a separate chamber in the ICU or in private room in the clinic.

Consent and recruitment procedures will be done in such a way that it will not be disclosed to other patients in the trauma room or in the ward. The information regarding patient's enrollment will be kept confidential and all study related interactions with the subject/patient's legal representative will be done in isolated room in the wards or in the clinics to maintain complete privacy. To safeguards the severe trauma patients, informed consent will be taken to participate in research by a legally authorized representative on behalf of a cognitively impaired subject. In absence of any legally authorized representative, the investigators will use emergency consent (Exception from Informed Consent Requirements for Emergency Research" Policy # 11026).

Patients who partially recover cognition will be asked to provide Assent and those fully recovered their cognition to understand the study will be asked for informed consent to continue participation. For trauma patients who are unconscious, under severe shock and are physically and mentally unfit to communicate, legally authorized representative will be identified with the help of patient's attendants. Explaining the consent will take around half an hour, and if the legal representative consented to allow subject participation within 5 hours of admission, he/she will be enrolled. Since the research investigations needs to be done during early hours of admission waiting time could be maximum 2-3 hours post admission. This study did not include any specific procedure which could provide distress to the participants. And the subject's privacy will be specifically taken care.

Sample size estimation: There is lack of information on the incidence of stress-induced hyperglycemia among trauma patients in Qatar. However, the current literature reported the incidence of stress-induced hyperglycemia (≥200 mg/dl) in trauma patients ranges from 10%-17% for all trauma admissions [3,4]. Therefore, taking the frequency of hyperglycemia to be 15% with 5% confidence limit and 97% confidence level, a total of 250 consecutive trauma patients needs to be included in the study. The investigators aim to complete the target of subject recruitment within 12 months and this research may take 18 months to be completed.

Bio-specimens: The blood specimen for research (10 ml initially after recruitment and 5 ml after 24 and 48 hours of admission) will be drawn together with the routine blood investigation.

For each study participant, blood will be drawn on admission to investigate Hemoglobin, HbA1C, blood glucose levels, Lactate, Base Deficit, High sensitive troponin T (HsTnT), Interleukin-6, Interleukin-18 and high sensitive C-reactive protein. Moreover, after 24 and 48 hours of admission, fasting blood glucose levels, hemoglobin, Lactate, Base Deficit, Interleukin-6, Interleukin-18 and high sensitive C-reactive protein will be repeated for all the patients. The main exposure will be hyperglycemia, defined as serum glucose 200 mg/dL or more. This level of glucose has previously been used by several trauma studies, and it is a commonly utilized cutoff to define hyperglycemia. Diabetes mellitus will be determined by patient history and/or admission HbA1c ≥ 6.5%. This level of HbA1c is based on current recommendations for the diagnosis of diabetes mellitus from the American Diabetes Association [10]. All the study participants will be managed according to the standard care of the hospital.

The investigators expect to enroll 250 consecutive trauma patients to be included in the study from the Hamad General Hospital, Doha, Qatar (this number of participants will be per center in case it becomes multicenter study to reach 750-1000 in total). The subject will be in the research until discharge from the hospital or died in the hospital and there will be no follow-up visits for the research.

Data collection & integrity: For each study participant, information will be collected regarding demographics (e.g., age, sex, nationality), injury (i.e., injury mechanism, ISS), and clinical characteristics (i.e., hospital stay, ICU days, and days on ventilator support). Information will be collected regarding outcomes, including mortality and in-hospital complications (i.e., pneumonia, renal failure, sepsis, Acute Respiratory Distress Syndrome and multiorgan failure).

The principal investigator (PI) will provide specific pre-assigned numbers to each sample collected and only the PI will know the subject identifier and all others will work with the number only. However, in the process of receiving and storage of samples, one appointed technical staff of laboratory services can have the access to the blood specimens. The investigator will track all the specimens received by allotting unique subject identifier for all blood specimens and track the sample transportation, processing, and consumption. Each sample will be labeled properly in color-coded cryo boxes at -80°C and will be discarded immediately after the test. Only the PI will have the access to the data which has been coded with subject identifier. The de-identified data from the individual data collection sheet will be entered by the research coordinator into the password protected Excel file.

Participation in this study is voluntary and the participant can be discontinued at any time, if he/she is willing to withdraw. If the participant is interested to withdraw from the study, he/she needs to contact the lead principle investigators of the study and this decision will not affect their medical care. In case of subjects recruited by emergency consent, after patient recovery he/she will have the right to withdraw from the study at any time voluntarily. If the patient chooses to withdraw from the study, they will be asked for permission to use their data up to the time of withdrawal. Data will be collected up to the time of withdrawal. Data will be collected up to the time of withdrawal. The existing data will not be removed from research and will be used for intention-to-treat analysis. However, the specimens will be discarded and no further data will be generated.

Data management: Data collection sheet will be used to record all relevant information of individual subjects. The de-identified data from the individual data collection sheet will be entered by the research coordinator into the password protected Excel file. Only the PI will have the access to the data which has been coded with subject identifier. The PI designated research team member will have the access to the de-identified data. Data will be stored and secured at logbook/secured computer with the PI. Hard copies will also be stored in closed envelopes in locked cabinets in PI's office. The data will be kept for a period of five years and then later will be destroyed. Data will be stored by the Hamad Trauma Center (HTC) Lead PI from all the participating centers and no data will be transferred from HTC to other centers. This study is opened for collaborative centers to be a multicenter study.

ELIGIBILITY:
Inclusion Criteria:

* All adult (≥18 years) male and female trauma patients consented for participation and have been investigated for random plasma glucose level and HbA1C measured within 5 hours of hospital admission will be included in the study.

Exclusion Criteria:

* Patients who descend to participate or in whom random serum glucose level and HbA1C not measured within 5 hours of hospital admission will be excluded from the study.
* Also, vulnerable populations (children, and pregnant women), and alcoholics will be excluded from the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult (≥18 years) trauma patients required hospital admission will be screened for participation in this study.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2016-10; Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
All cause Mortality | 30 days

SECONDARY OUTCOMES:
Pneumonia | 30 days
  ventilator acquired infection
Sepsis | 30 days
  The new definitions published in Journal of American Medical Association (2016;315:801-810)
Multiorgan failure | 30 days
Hospital length of stay | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Ayman El-Menyar, MD, Principal Investigator — Hamad Medical Coorporation
Locations (1):
- Hamad Medical Coorporation, Doha, Qatar

IPD SHARING:
Plan to Share IPD: No
Only the lead PI will have the access to the data which will be coded with subject identifier to ensure data safety and confidentiality. The study will be opened for collaboration with multi-centers. Data from other centers will be shared with the Lead PI.

REFERENCES:
- [Background] McCowen KC, Malhotra A, Bistrian BR. Stress-induced hyperglycemia. Crit Care Clin. 2001 Jan;17(1):107-24. doi: 10.1016/s0749-0704(05)70154-8. PMID 11219223
- [Background] Yendamuri S, Fulda GJ, Tinkoff GH. Admission hyperglycemia as a prognostic indicator in trauma. J Trauma. 2003 Jul;55(1):33-8. doi: 10.1097/01.TA.0000074434.39928.72. PMID 12855878
- [Background] Laird AM, Miller PR, Kilgo PD, Meredith JW, Chang MC. Relationship of early hyperglycemia to mortality in trauma patients. J Trauma. 2004 May;56(5):1058-62. doi: 10.1097/01.ta.0000123267.39011.9f. PMID 15179246
- [Background] Kerby JD, Griffin RL, MacLennan P, Rue LW 3rd. Stress-induced hyperglycemia, not diabetic hyperglycemia, is associated with higher mortality in trauma. Ann Surg. 2012 Sep;256(3):446-52. doi: 10.1097/SLA.0b013e3182654549. PMID 22868366
- [Background] Bosarge PL, Shoultz TH, Griffin RL, Kerby JD. Stress-induced hyperglycemia is associated with higher mortality in severe traumatic brain injury. J Trauma Acute Care Surg. 2015 Aug;79(2):289-94. doi: 10.1097/TA.0000000000000716. PMID 26218699
- [Background] Rovlias A, Kotsou S. The influence of hyperglycemia on neurological outcome in patients with severe head injury. Neurosurgery. 2000 Feb;46(2):335-42; discussion 342-3. doi: 10.1097/00006123-200002000-00015. PMID 10690722
- [Background] Wei Y, Chen K, Whaley-Connell AT, Stump CS, Ibdah JA, Sowers JR. Skeletal muscle insulin resistance: role of inflammatory cytokines and reactive oxygen species. Am J Physiol Regul Integr Comp Physiol. 2008 Mar;294(3):R673-80. doi: 10.1152/ajpregu.00561.2007. Epub 2007 Dec 19. PMID 18094066
- [Background] Esposito K, Marfella R, Giugliano D. Plasma interleukin-18 concentrations are elevated in type 2 diabetes. Diabetes Care. 2004 Jan;27(1):272. doi: 10.2337/diacare.27.1.272. No abstract available. PMID 14694002
- [Background] Dungan KM, Braithwaite SS, Preiser JC. Stress hyperglycaemia. Lancet. 2009 May 23;373(9677):1798-807. doi: 10.1016/S0140-6736(09)60553-5. PMID 19465235
- [Derived] El-Menyar A, Asim M, Mir F, Hakim S, Kanbar A, Siddiqui T, Younis B, Ahmed K, Mahmood I, Atique S, Al Jogol H, Taha I, Mustafa F, Alabdallat M, Abdelrahman H, Peralta R, Al-Thani H. Patterns and Effects of Admission Hyperglycemia and Inflammatory Response in Trauma Patients: A Prospective Clinical Study. World J Surg. 2021 Sep;45(9):2670-2681. doi: 10.1007/s00268-021-06190-5. Epub 2021 Jun 11. PMID 34117510